CLINICAL TRIAL: NCT05946967
Title: Colon Transit Study for Assessment of Chronic Constipation and Therapy Directed Against Fecal Evacuation Disorder by Biofeedback With or Without Transcutaneous Electrical Stimulation of Posterior Tibial Nerve
Brief Title: Colon Transit Study for Chronic Constipation Assessment and Therapy by Biofeedback With and Without TENS
Acronym: TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-128-DM-131
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Constipation
Keywords: CTT; IBS-C; Functional-constipation
MeSH Terms: conditions — Constipation | interventions — Biofeedback, Psychology; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofeedback with TENS (Active Comparator): Patients with constipation will undergo biofeedback treatment along with transcutaneous electrical stimulation (TENS)
  Interventions: Other: Biofeedback with TENS
- Biofeedback only (Sham Comparator): Patients with constipation will undergo biofeedback treatment only
  Interventions: Other: Biofeedback only

INTERVENTIONS:
Other: Biofeedback with TENS — Constipation patients will be given biofeedback treatment along with transcutaneous electrical stimulation (TENS) of posterior tibial nerve
  Arms: Biofeedback with TENS
Other: Biofeedback only — Constipation patients will be given biofeedback treatment only
  Arms: Biofeedback only

SUMMARY:
One of the most challenging functional gastrointestinal illnesses (FGID) to manage is constipation, which is a widespread issue. The fact that constipation can be caused by a variety of conditions, including slow colon transit, faecal evacuation disorder, or a combination of both slow colon transit and faecal evacuation disorder, is one of the main reasons it is challenging to treat. Treatment options vary based on the pathogenetic mechanism; for instance, biofeedback, botulinum toxin injections in the puborectal sling, or transcutaneous electrical nerve stimulation (TENS) are required to treat faecal evacuation problem. On the other hand, prucalopride and other colokinetic drugs as well as drugs that promote high amplitude propagating contractions, including bisacodyl and sodium pyrosulphate, are used to treat slow transit constipation. Sometimes faecal evacuation disorders that inhibit the evacuation of the transit markers can cause slow colon transit times; these secondary sluggish colon transit times have been shown to improve with biofeedback therapy alone. Even though the causes of faecal evacuation disorders are not fully understood, it is known that abnormal neuromuscular function is the result. A few workers have stimulated the posterior tibial nerve, another sacral plexus branch, non-invasively with TENS. Studies on the use of biofeedback in the treatment of patients with faecal evacuation problems are lacking. Accordingly, we wish to undertake a prospective study with following aims: (i) To assess safety and efficacy of colon transit study by an indigenous radio opaque marker to identify the mechanism of constipation and to assess outcome of treatment (improvement of transit time). (ii) To assess the efficacy of pathogenesisdirected therapy such as biofeedback with or without TENS for posterior tibial nerve to treat fecal evacuation disorder. (iii) To assess colon transit following treatment of fecal evacuation disorder with either biofeedback alone or biofeedback with TENS for posterior tibial nerve.

DETAILED DESCRIPTION:
Introduction Constipation is a common problem and one of the most difficult functional gastrointestinal diseases (FGID) to treat. An Asian survey showed that among patients with FGID, constipation patients are most dissatisfied with treatment . One of the major reasons why constipation is difficult to treat is because of the fact that constipation may result from multiple factors like slow colon transit, fecal evacuation disorder, or a combination of both slow colon transit and fecal evacuation disorder . Until and unless the exact cause is identified, the empirical treatment with laxatives does not work. Treatment varies depending upon the pathogenetic mechanism, for example, fecal evacuation disorder needs to be treated with biofeedback , botulinum toxin injection in the puborectal sling, or transcutaneous electrical nerve stimulation (TENS) . On the other hand, slow transit constipation is treated with colokinetic agents such as prucalopride and agents stimulating high amplitude propagated contractions such as bisacodyl and sodium pyrosulphate. Sometimes colon transit time may be slow secondary to fecal evacuation disorder mitigating evacuation of the transit markers; such secondary slow colon transit has been shown to improve with biofeedback therapy alone.

Fecal evacuation disorders are diagnosed with anorectal manometry, balloon expulsion test, and barium or magnetic resonance imaging defecography. On the other hand, slow transit constipation is diagnosed by radio-nuclide colon transit study, a colon transit study using radio-opaque markers and smart pills, etc. Since these investigations are not widely available, it becomes difficult to detect the mechanism of constipation in practice by many physicians and gastroenterologists. Two tests that can be easily performed in office practice by most physicians and gastroenterologists include: (i) balloon expulsion test, (ii) colon transit time (CTT) by opaque markers. Detecting these pathophysiological mechanisms of chronic constipation is expected to provide personalized therapy for these patients.

Though mechanisms of fecal evacuation disorders are poorly understood, yet it is known that it results from abnormal neuromuscular function resulting in lack of increase in intra-rectal pressure during attempted defecation and failure of relaxation of pelvic floor muscles. This led to some workers to treat these patients with sacral nerve stimulation, which is primarily used to treat fecal incontinence. However, sacral nerve stimulation is quite invasive, requires major surgical procedure and is associated with multiple complications, including infection. A few workers have used non-invasive TENS to stimulate posterior tibial nerve, which is also a branch of sacral plexus. However, there is lack of studies to treat patients with fecal evacuation disorders with or without biofeedback, which is considered, the first-line therapy for fecal evacuation disorder. Accordingly, we hypothesized that, (i) the office-based investigation such as colon transit study using radio-opaque markers will be useful to diagnose fecal evacuation disorder, which will be able to direct further therapy, (ii) biofeedback with TENS for posterior tibial nerve will be superior to biofeedback alone to treat fecal evacuation disorder, and (iii) successful treatment of fecal evacuation disorder with either biofeedback alone or biofeedback with TENS for posterior tibial nerve will improve colon transit as assessed by radio-opaque marker study.

Accordingly, we wish to undertake a prospective study with following aims:

(i) To assess safety and efficacy of colon transit study by an indigenous radio opaque marker to identify the mechanism of constipation and to assess outcome of treatment (improvement of transit time).

(ii) To assess the efficacy of pathogenesis-directed therapy such as biofeedback with or without TENS for posterior tibial nerve to treat fecal evacuation disorder.

(iii) To assess colon transit following treatment of fecal evacuation disorder with either biofeedback alone or biofeedback with TENS for posterior tibial nerve.

Methodology

Inclusion criteria:

i) Patient with refractory chronic constipation ii) >18 years of age Exclusion criteria i) Patient with uncontrolled diabetes/ untreated thyroid/ organic disease ii) No lower limb iii) <18 years of age

Fifty patients with chronic constipation will undergo the below-mentioned tests as per standardized protocol. It is important to mention here that all these tests are standard of care for these patients. The tests are: (i) anorectal manometry, (ii) balloon expulsion, (iii) colon transit study by an indigenous radio-opaque marker according to the standard of care, and (iv) defecography (either barium or magnetic resonance imaging).

The diagnostic criteria for fecal evacuation disorder will be as follows: positive result in 2 of the following tests - a) anorectal manometry with defecation index of <1.4, b) abnormal balloon expulsion test, c) abnormal defecography.

The ability of CTT to diagnose fecal evacuation disorder and slow transit constipation among these subjects will be assessed. Patients with fecal evacuation disorders diagnosed as above will be subjected to daily biofeedback with one group receiving TENS daily and the other group receiving sham stimulations. These treatments will be given for 10 days. The treatment group shall be decided based upon the understanding with patients and mutual decision of the doctor and the patient. Standard treatment of stimulative laxatives will be given to patients with bloating and ispaghula husk to patients without bloating.

No patient will have to pay for biofeedback and TENS. The other tests (anorectal manometry, balloon expulsion, colon transit study, and defecography) are standard of care for patients with constipation. Follow up will be done at 1 month and 3 months as described in figure 2.

Outcome measures i) Constipation severity questionnaire will be used to assess the Constipation Scoring System.

ii) Number of spontaneous bowel movements, time spent in the toilet, stool form (according to Bristol stool chart) will be assessed with a stool diary.

iii) Dose of laxatives used. iv) After the end of treatment, colon transit study will be repeated to assess its improvement.

ELIGIBILITY:
Inclusion Criteria:

* i) Patient with refractory chronic constipation ii) 18-65 years of age

Exclusion Criteria:

* i) Patient with uncontrolled diabetes/ untreated thyroid/ organic disease ii) No lower limb iii) <18 years of age iv) >65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Constipation severity | 3 months
  Constipation severity questionnaire will be used to assess the Constipation Scoring System
Bowel movement assessment | 3 months
  Number of spontaneous bowel movements, time spent in the toilet, stool form (according to Bristol stool chart) will be assessed with a stool diary
Treatment effect | 3 months
  After the end of treatment, colon transit study will be repeated to assess its improvement.

SECONDARY OUTCOMES:
Dose of laxatives | 3 month
  Dose of laxatives used will be recorded